CLINICAL TRIAL: NCT06571578
Title: High Intensity Interval Inspiratory Training Effect on Ventilatory Functions and Diaphragmatic Excursion in Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Abd el Maboud Youssef, assisstant lecture, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMT for FHS
Record Dates: First submitted 2024-08-13; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: FHD

STUDY DESIGN:
Intervention Model Description: randomised control trial (RCT)
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exoerimental Group (Experimental): Thirty subjects will receive combined program containing interval inspiratory muscle training and conventional exercise program for FHP 12 weeks (3 sessions/ week).
  Interventions: Device: Threshold Inspiratory muscle trainer; Other: posture correction exercises
- Control Group (Other): control group Thirty subjects will receive a conventional exercise program for FHP for 12 weeks (3 sessions/ week).
  Interventions: Other: posture correction exercises

INTERVENTIONS:
Device: Threshold Inspiratory muscle trainer — threshold inspiratory muscle trainer device Each subject will breathe through a separate mouthpiece through attach the mouthpiece firmly While putting a nose clip and inhale deeply through the mouthpiece to generate an inspiratory pressure greater than the indicated presetting threshold pressure to compress the spring and open the valve. Using High - intensity interval training technique
  Other Names: posture correction exercises
  Arms: exoerimental Group
Other: posture correction exercises — conventional exercise consists of
  * Cervical isometric exercises will be performed in the sitting position by resisting at the forehead (cervical ﬂexion, extension, rotation and side bending) for 10 seconds with 15 seconds breaks between holds with 10-15 repetitions in a progressive manner 3time/week for 12 weeks.
  * Postural correction exercise consists of gently rolling of pelvis forward to an upright neutral sitting position, followed by scapular correction and occipital lift. Also, for the sub-occipital muscles stretching
  * stretching exercises for scalene and levator muscles

SUMMARY:
PURPOSE: ……… The purpose of the study is to investigate the effect of interval inspiratory muscle training on respiratory functions in subjects with forward head posture associated with chronic nonspecific neck pain

BACKGROUND: Alteration of head and neck positions can have an immediate negative effect on respiratory function. Clinicians should be prompted to assess respiratory function when assessing individuals with FHP and decrease the tension on respiratory system to avoid consequence. Also FHP has a negative effect on chest expansion and diaphragmatic function

the incidence of forward head posture increases nowadays due to increase using of smartphones HYPOTHESES:: There will be no a significant effect of interval inspiratory muscle training on respiratory functions in chronic forward head posture subjects.

RESEARCH QUESTION: Will the interval inspiratory muscle training improve respiratory functions in subjects forward head posture associated with chronic nonspecific neck pain?

DETAILED DESCRIPTION:
* For evaluation: we will assess 1-diaphragmatic excursion using ultrasonography 2- ventilatory functions using spirometer 3- chest expansion using tape measurement 4- height and weight scale to detect BMI 5- Craniocervical angle
* For treatment: we will use 1- threshold inspiratory muscle trainer

And they will be randomly allocated into two groups:

Experimental Group: Thirty subjects will receive combined program containing interval inspiratory muscle training and conventional exercise program for FHP 12 weeks (3 sessions/ week)

Control Group : Twenty subjects will receive conventional exercise program for FHP 12 weeks (3 sessions/ week)

ELIGIBILITY:
Inclusion Criteria:

* Sixty subjects (female) have forward heads and Their craniocervical angle is from 30 to 50°
* Their body mass index ranged from (24.9 -29.9) kg/m2

Exclusion Criteria:

* Chest diseases (either obstructive or restrictive).
* Smoker patient.
* Clinical signs of a severe cardiac event. (eg, congestive heart failure),
* Neurological disorders affecting respiratory muscles or any muscular dystrophies (cervical disc or bulge).
* Patient with haemodynamic instability.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female subjects from 18 to 25 years old with FHP
Enrollment: 60 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
improve ventilatory functions | 3 months
  measure ventilatory functions in percentage from predictied using spirometery (Digital-CONTEC-SP10-Spirometer-Lung Breathing-Diagnostic (Made in China), to measure ventilatory function test parameters.changes
  * Forced expiratory volume in the first second (FEV1)
  * Forced vital capacity (FVC).
  * FEV1/FVC ratio
  * Peak expiratory flow rate (PEFR).
Diaphragmatic execursion | 3 months
  Diaphragmatic sonography model (LOG IQ E10S) for measuring diaphragmatic excursion changes.in centimeter
chest expansion tests | 3 months
  Using tape Measurement tool: To measure chest expansion changes in centimetres at the suprasternal notch, at the nipple and xiphoid levels.

SECONDARY OUTCOMES:
craniocervical angle | 3 months
  • Markings were done with help of Kinovea software. The intersection of a horizontal line passing through C7 spinous process and line joining the midpoint of tragus of ear is known as Craniovertebral angle.
Body mass index | 3 months
  measuring body mass index kg\m2 before measuring ventilatory function test by measuring height in centimetres and body weight in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt